CLINICAL TRIAL: NCT01989078
Title: Losartan Treatment for Sickle Cell Chronic Kidney Disease
Brief Title: Losartan for Sickle Cell Kidney Disease
Acronym: SCD-Losartan
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Marianne Yee, MD, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00056125
Record Dates: First submitted 2013-02-26; First posted 2013-11-20 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Sickle Cell Disease
Keywords: Kidney disorder; Blood disorder; Pediatrics
MeSH Terms: conditions — Anemia, Sickle Cell; Kidney Diseases; Hematologic Diseases | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: Participants will all receive the study medication in addition to the standard of care treatment. There is no control group for this pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Losartan (Experimental): Participants taking losartan, in addition to taking hydroxyurea therapy, as prescribed per standard of care
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — Adults and Children >50 kg:
  * Those with systolic blood pressure (SBP) ≥ 100 mm Hg at entry will start with 50 mg of oral losartan once daily. At the week 2 visit, losartan will be increased to 100 mg daily.
  * Those with SBP <100 mm Hg at entry will start with 25 mg of oral losartan once daily. Participants will return after 1 week for titration to 50 mg daily, if tolerated (i.e. SBP not lower than pre-losartan measurement by 10 mm Hg or more), and after 2 weeks to monitor blood pressure.
  Children <50 kg weight:
  * Treatment will start with 25 mg oral Losartan once daily given as a morning dose. At the 2 week visit, Losartan will be increased to 50 mg daily. The dose will be increased to 100 mg once a body weight of 50 kg is achieved.
  Other Names: Cozaar

SUMMARY:
Sickle cell nephropathy (SCN) is a progressive complication of sickle cell disease (SCD) that begins in childhood and results in renal (kidney) failure and early mortality in nearly 12% of adults with hemoglobin SS (HbSS). The potential for prevention and reversal of kidney damage in SCD is not known. Albuminuria is a commonly used biomarker of glomerular damage; however the correlations of albuminuria with specific measurements of glomerular function and pathophysiology have not been determined. The investigators hypothesize that in patients with persistent albuminuria despite treatment of SCD with hydroxyurea, losartan will reverse kidney dysfunction in early stage nephropathy and ameliorate progressive kidney dysfunction in more advanced nephropathy. The primary aim is to study the acute and longer-term effects of losartan (study drug) on specific glomerular functions in children and adults with SCD who have persistent albuminuria. Research glomerular function tests will be done at study entry (prior to taking losartan), 1 month, and 1 to 2 years after starting losartan therapy (participants may take losartan for up to 24 months). In addition, participants are seen each month in clinic and assessed by their regular clinical team. The second aim is to assess the correlation of changes in albuminuria after 1 month of losartan with changes in direct measurements of glomerular function at 12-24 months, thus determining if the magnitude of the initial decrease in albuminuria in response to losartan predicts sustained improvements in renal function.

DETAILED DESCRIPTION:
Sickle cell nephropathy (SCN) is a progressive complication of sickle cell disease (SCD) that begins in childhood and results in renal (kidney) failure and early mortality in nearly 12% of adults with hemoglobin SS (HbSS). The potential for prevention and reversal of kidney damage in SCD is not known. Albuminuria is a commonly used biomarker of glomerular damage; however the correlations of albuminuria with specific measurements of glomerular function and pathophysiology have not been determined. The investigators hypothesize that in patients with persistent albuminuria despite treatment of SCD with hydroxyurea, losartan will reverse kidney dysfunction in early stage nephropathy and ameliorate progressive kidney dysfunction in more advanced nephropathy. Losartan is an FDA-approved drug to treat blood pressure to protect the kidneys in people who have diseases like diabetes and blood pressure. It is not specifically labeled for use in sickle cell disease. Participants will be enrolled from Children's Healthcare of Atlanta (pediatric subjects) or Grady Memorial Hospital (adult subjects) and will be in the study for 1 to 2 years (depending on when the final renal function tests can be preformed).

The primary aim of this pilot study is to evaluate the acute and longer-term effects of losartan (study drug) on renal function in children and adults with SCD who have persistent albuminuria. The renal function tests will be done at study entry (prior to taking losartan), 1 month, and 1 to 2 years after starting losartan therapy. In addition, participants are assessed monthly by their regular clinical team. The second aim of this study is to assess the correlation of changes in albuminuria after 1 month of losartan with changes in direct measurements of renal function at 12-24 months, thus determining if the magnitude of the initial decrease in albuminuria in response to losartan predicts sustained improvements in renal function.

ELIGIBILITY:
Inclusion Criteria:

* SCD genotype HbSS or HbS/beta-0-thalassemia
* Age greater than or equal to 9 years old
* Urinary albumin/creatinine ratio (ACR) greater than or equal to 30 mg/gram creatinine on greater than or equal to 2 occasions separated by one month or more
* Current treatment with hydroxyurea and a sustained hematologic response for 6 months or more prior to enrollment

Exclusion Criteria:

* End-stage renal failure (estimated GFR <30 ml/min/1.73 m2)
* Known co-existent medical conditions that could affect the kidneys, such as diabetes mellitus, systemic lupus erythematosus (SLE), or human immunodeficiency virus (HIV) positive
* Chronic therapy (daily use for ≥8 weeks) with non-steroidal anti-inflammatory drugs (NSAIDs)
* Females who are pregnant
* Pre-existing hyperkalemia (serum potassium > 5.5 milliequivalents per liter (mEq/L))
* Current chronic transfusion therapy

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in albumin/creatinine ratio (ACR) | Baseline, Month 1, End of treatment (12 to 24 months)
  The effects of losartan on the mean change in albumin/creatinine ratio (ACR) will be examined.
Change in glomerular filtration rate (GFR) | Baseline, Month 1, End of treatment (12 to 24 months)
  The effects of losartan on the mean change in glomerular filtration rate (GFR) will be examined.
Change in renal plasma flow (RPF) | Baseline, Month 1, End of treatment (12 to 24 months)
  The effects of losartan on the mean change in renal plasma flow (RPF) will be examined.
Change in glomerular permeability (GP) | Baseline, Month 1, End of treatment (12 to 24 months)
  The effects of losartan on the mean change in glomerular permeability (GP) will be examined.

OTHER OUTCOMES:
Association between changes in albumin/creatinine ratio (ACR) at one month and glomerular filtration rate (GFR) at 12 months | Baseline, Month 1, End of treatment (12 to 24 months)
  For the exploratory aims, the relationship between the degree of short-term change in albumin/creatinine ratio (ACR) and longer-term changes in glomerular filtration rate (GFR) will be examined. The mean change in urinary ACR after 1 month of treatment with losartan will be associated with the long-term mean changes in GFR after 12 months of treatment.
Association between changes in albumin/creatinine ratio (ACR) at one month and renal plasma flow (RPF) at 12 months | Baseline, Month 1, End of treatment (12 to 24 months)
  For the exploratory aims, the relationship between the degree of short-term change in albumin/creatinine ratio (ACR) and longer-term changes in renal plasma flow (RPF) will be examined. The mean change in urinary ACR after 1 month of treatment with losartan will be associated with the long-term mean changes in RPF after 12 months of treatment.
Association between changes in albumin/creatinine ratio (ACR) at one month and glomerular permeability (GP) at 12 months | Baseline, Month 1, End of treatment (12 to 24 months)
  For the exploratory aims, the relationship between the degree of short-term change in albumin/creatinine ratio (ACR) and longer-term changes in glomerular permeability (GP) will be examined. The mean change in urinary ACR after 1 month of treatment with losartan will be associated with the long-term mean changes in GP after 12 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Yee, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health Systems, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia